CLINICAL TRIAL: NCT03515694
Title: Minimal Optimal Dose of Sugammadex in Elective Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRIDION_ERASME
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-04

CONDITIONS: Time of a TOF Ratio >0,9
Keywords: Bridion; Sugammadex; TOF
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: Parallel, Double blind Monocentric Prospective Vs placebo
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Dose of 0mg/kg TOF1 (Placebo Comparator)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 0mg/kg TOF2 (Placebo Comparator)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 0 ,5mg/kg TOF1 (Experimental)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 0,5mg/kg TOF2 (Active Comparator)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 1mg/kg TOF1 (Experimental)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 1mg/kg TOF2 (Active Comparator)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 2mg/kg TOF1 (Experimental)
  Interventions: Drug: Sugammadex Injection [Bridion]
- Dose of 2mg/kg TOF2 (Active Comparator)
  Interventions: Drug: Sugammadex Injection [Bridion]

INTERVENTIONS:
Drug: Sugammadex Injection [Bridion] — Injection of 10mL of translucide solution

SUMMARY:
Time of appearance of TOF Ratio >0,9 with different doses of Sugammadex

DETAILED DESCRIPTION:
Design: monocentric, prospective, controlled, randomized, double-blind study Inclusion criteria: women and men> 18 years old, elective surgery, BMI <30, patients giving consent to free and informed participation in writing;

Exclusion criteria:

* minor patients;
* Patients refusing to sign the consent;
* Patients included in another protocol within 3 months;
* Pregnant or lactating patients;
* Patients with a history of allergy to Sugammadex;
* Patients with known neuromuscular disease;
* Patients with renal or hepatic impairment.

Course of the study :

* 40 patients will be recruited at the time of the anesthesia consultation and randomized to double blind in 8 groups (the day before surgery)
* All patients will benefit from general anesthesia. Anesthetic management

  (1- 3mg / kg / IV propofol, 0.2 μg / IV sufentanil, 0.6 mg / kg rocuronium and maintenance anesthesia with sevoflurane) will be standardized for all patients.
* Upon administration of rocuronium the acceleromyography transducer will be attached to the distal phalanx of the thumb, and repeated TOF stimulation will be applied to the ulnar nerve wrist at intervals of 15 seconds. Neuromuscular monitoring is continued until the end of the anesthesia.
* Once the first answer (1st twitch) appeared a dose of sugammadex will be administered according to the group whose patient was randomized: Test Groups Control Groups Group 1: Placebo + TOF 1 Group 1bis: Placebo + TOF2 Group 2: 0.5 mg / kg + TOF1 Group 2bis: 0.5 mg / kg + TOF2 Group 3: 1mg / kg + TOF1 Group 3bis: 1mg / kg + TOF2 Group 4: 2mg / kg + TOF 1 Group 4bis: 2mg / kg + TOF 2
* Then a standard dose of 4mg / kg will be administered at the end of the procedure before awakening to all patients who have signs of residual curarization (TOF ratio <0.9). The pharmacy will be responsible for preparing the different doses of sugammadex, the syringe will be carefully covered and packaged, will contain an equal volume so that the anesthetists do not know which group the patient belongs to. Data collection: In real time during the intervention by the anesthesiologist in charge of patient Method of Analysis: Analysis of intent-to-treat data

ELIGIBILITY:
Inclusion Criteria:

women and men> 18 years of age Elective Surgery BMI <30, patients who gave consent to free and informed participation in writing

Exclusion Criteria:

* minor patients;
* patients refusing to sign consent;
* patients included in another protocol within 3 months;
* pregnant or nursing patients;
* patients with a history of allergy to Sugammadex;
* patients with known neuromuscular disease
* patients with renal or hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the recovery time of the ratio 0.9. | 1 hour
  Evaluate the recovery time of the ratio 0.9.

SECONDARY OUTCOMES:
Time of appearance of 4 responses to the TOF | 1 hour
  Time of appearance of 4 responses to the TOF
Evaluate the four-to-four ratio <0.7 after total recovery. | 1 hour
  Evaluate the four-to-four ratio <0.7 after total recovery.
Watch time at the recovery room. | 4 hours
  Watch time at the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy FERNANDEZ, Resident, Principal Investigator — Erasme University Hospital
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided